CLINICAL TRIAL: NCT02681094
Title: A Multi-Center, Randomized, Double-Blind, Active-Controlled , Parallel Group, Phase III Trial to Evaluate the Safety and Efficacy of Saxagliptin 5mg Co-administered With Dapagliflozin 5mg Compared to Saxagliptin 5mg or Dapagliflozin 5mg All Given as Add-on Therapy to Metformin inPatients With Type 2 Diabetes Who Have Inadequate Glycaemic Control on Metformin Alone
Brief Title: A Multi-Center, Randomized, Double-Blind, Phase III Trial to Evaluate the Safety and Efficacy of Saxagliptin Co-administered With Dapagliflozin Compared to Saxagliptin or Dapagliflozin All Given as add-on Therapy to Metformin in Subject With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D1683C00005
Record Dates: First submitted 2016-02-10; First posted 2016-02-12 (Estimated); Results first posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-09

CONDITIONS: Type 2 Diabetes Mellitus; Inadequate Glycaemic Control
Keywords: Diabetes Mellitus Type 2,; saxagliptin,; dapagliflozin,; metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; saxagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Saxagliptin+Dapagliflozin+Metformin (Active Comparator): 5 mg Tablets, Oral, Once daily, 24 weeks for Saxagliptin and Dapagliflozin
  Interventions: Drug: Dapagliflozin; Drug: Saxagliptin
- Dapagliflozin+Saxagliptin placebo+Metformin (Active Comparator): 5 mg Tablets, Oral, Once daily, 24 weeks for Dapagliflozin and Saxagliptin Placebo
  Interventions: Drug: Dapagliflozin; Drug: Placebo for Saxagliptin
- Saxagliptin+Dapagliflozin placebo+metformin (Active Comparator): 5 mg Tablets, Oral, Once daily, 24 weeks for Saxagliptin and Dapagliflozin placebo
  Interventions: Drug: Placebo for Dapagliflozin; Drug: Saxagliptin

INTERVENTIONS:
Drug: Dapagliflozin — 5mg, orally, Green, plain, diamond-shaped, film-coated tablet
  Other Names: Forxiga
  Arms: Dapagliflozin+Saxagliptin placebo+Metformin; Saxagliptin+Dapagliflozin+Metformin
Drug: Placebo for Dapagliflozin — Does not contain active ingredient, orally, Green, plain, diamond-shaped, film-coated tablet
  Arms: Saxagliptin+Dapagliflozin placebo+metformin
Drug: Saxagliptin — 5mg, orally, Plain, yellow, biconvex, round, film-coated tablet
  Other Names: Onglyza™
  Arms: Saxagliptin+Dapagliflozin placebo+metformin; Saxagliptin+Dapagliflozin+Metformin
Drug: Placebo for Saxagliptin — Does not contain active ingredient, orally, Plain, yellow, biconvex, round, film-coated tablet
  Arms: Dapagliflozin+Saxagliptin placebo+Metformin

SUMMARY:
The aim of this study is to evaluate safety and efficacy of therapy with saxagliptin 5mg co-administered with dapagliflozin 5mg, compared to therapy with saxagliptin 5mg or dapagliflozin 5mg in patients who are inadequately controlled on ≥1500mg/day of metformin monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years old at time of informed consent;
2. Patients with Type 2 diabetes mellitus (T2DM) defined as HbA1C≥7.5% to ≤10.0% at screening visit;
3. Stable metformin therapy for at least 8 weeks prior to enrolment at a dose of ≥1500mg per day;
4. BMI ≤45.0kg/m2 at Enrolment visit;
5. Fasting Plasma Glucose (FPG) ≤ 270mg/dl(15.0mmol/L) at the enrolment visit;
6. For Females Only: Women of childbearing potential (WOCBP) must be using an acceptable method of contraception to avoid pregnancy throughout the study and for at least 4 weeks after the last dose of study medication in such a manner that the risk of pregnancy is minimized.

Exclusion Criteria:

1. History of diabetes insipidus, Type 1 diabetes or Latent Autoimmune Diabetes of Adults, diabetic ketoacidosis or hyperosmolar nonketotic coma and Symptoms of poorly controlled diabetes that would preclude participation in this trial including but not limited to marked polyuria and polydipsia with greater than 10% weight loss during the 3 months prior to Enrolment (Visit 1), or other signs and symptoms.
2. History of pancreatitis.
3. Administration of any antihyperglycaemic therapy, other than metformin, for more than 14 days (consecutive or not) during the 8 weeks prior to enrolment
4. Any use of DPP-4 inhibitor or SGLT-2 inhibitor within 8 weeks prior to enrolment.
5. Significant hepatic disease, including, but not limited to, chronic active hepatitis and/or severe hepatic insufficiency and/or significant abnormal liver function, including patients with Alanine transaminase (ALT) and/or Aspartate transaminase (AST) ≥3x ULN (Upper Limit of Normal)and/or Total Bilirubin ≥2.0x ULN. History of severe hepatobiliary disease or hepatotoxicity with any medication. Positive serologic evidence of current infectious liver disease, including patients who are known to be positive for Hepatitis viral antibody ImmunoglobulinM (IgM), Hepatitis B surface antigen, and Hepatitis C virus antibody.
6. Moderate or severe impairment of renal function [defined as Estimated Glomerular Filtration Rate (eGFR) <60milliLitre/min/1.73 m2 (estimated by Modification in Diet and Renal Disease (MDRD)) or serum creatinine ≥1.5mg/dL in males or ≥1.4mg/dL in females]. Conditions of congenital renal glucosuria, history of unstable or rapidly progressing renal disease.
7. History of any clinically significant disease or disorder which, in the opinion of the investigator, may put the patient at risk because of participation in the study, may influence the results, or may limit the patient's ability to participate in or complete the study.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 905 (Actual)
Dates: Start 2016-02-26 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (95):
- United States (44):
  - Research Site, Saraland, Alabama
  - Research Site, Fresno, California
  - Research Site, Harbor City, California
  - Research Site, Hawaiian Gardens, California
  - Research Site, Lancaster, California
  - Research Site, Los Angeles, California
  - Research Site, Montclair, California
  - Research Site, Pomona, California
  - Research Site, Spring Valley, California
  - Research Site, Vallejo, California
  - Research Site, Denver, Colorado
  - Research Site, Northglenn, Colorado
  - Research Site, Wheat Ridge, Colorado
  - Research Site, Waterbury, Connecticut
  - Research Site, Cooper City, Florida
  - Research Site, Doral, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Buford, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Hazel Crest, Illinois
  - Research Site, New Orleans, Louisiana
  - Research Site, Zachary, Louisiana
  - Research Site, Biloxi, Mississippi
  - Research Site, Florissant, Missouri
  - Research Site, Albany, New York
  - Research Site, The Bronx, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Mooresville, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Columbus, Ohio
  - Research Site, Maumee, Ohio
  - Research Site, East Providence, Rhode Island
  - Research Site, West Columbia, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Odessa, Texas
  - Research Site, Sugar Land, Texas
  - Research Site, Waco, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Norfolk, Virginia
- Canada (13):
  - Research Site, Moncton, New Brunswick
  - Research Site, Bridgewater, Nova Scotia
  - Research Site, Brampton, Ontario
  - Research Site, Etobicoke, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, London, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Lévis, Quebec
  - Research Site, Mirabel, Quebec
  - Research Site, Pointe-Claire, Quebec
  - Research Site, Saint-Marc-des-Carrieres, Quebec
- Czechia (9):
  - Research Site, Chrudim III
  - Research Site, České Budějovice
  - Research Site, Jílové u Prahy
  - Research Site, Ostrava
  - Research Site, Pardubice
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Praha Klanovice
  - Research Site, Uherské Hradiště
- Germany (14):
  - Research Site, Berlin
  - Research Site, Bünde
  - Research Site, Essen
  - Research Site, Giengen an der Brenz
  - Research Site, Großheirath
  - Research Site, Hof
  - Research Site, Hohenmölsen
  - Research Site, Karlsruhe
  - Research Site, Lichtenfels
  - Research Site, Meine
  - Research Site, Münster
  - Research Site, Rehburg-Loccum
  - Research Site, Stolberg
  - Research Site, Villingen-Schwenningen
- Mexico (4):
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, Zapopan
- Russia (11):
  - Research Site, Arkhangelsk
  - Research Site, Izhevsk
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Perm
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Tver'
  - Research Site, Ufa
  - Research Site, Vladikavkaz
  - Research Site, Yekaterinburg

REFERENCES:
- See also: d1683c00005 csp Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3863&filename=d1683c00005_csp_Redacted.pdf
- See also: D1683C00005 SAP redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3863&filename=D1683C00005_SAP_redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 119 sites in 6 countries: Canada, Czech Republic, Germany, Mexico, Russia, and United States (US). Approximately 900 participants were to be randomized. Participants with Type 2 Diabetes (T2DM) inadequately controlled on metformin alone were randomized in this study.
Pre-assignment Details: All participants had screening (Visit 0) at 1 week prior to enrolment to screen the eligibility based on non-fasting sample of Glycated haemoglobin (Hb A1c); results of HbA1c determined enrolment based on inclusion/exclusion criteria. An abbreviated informed consent was signed and review of concomitant or other medications/therapies were performed.
Groups:
- Dapagliflozin + Saxagliptin + Metformin: Randomized participants received orally once daily (QD) dapagliflozin 5 mg and saxagliptin 5 mg film coated tablets as an add-on to metformin (≥1500 mg/day orally)
- Dapagliflozin + Metformin: Randomized participants received orally QD dapagliflozin 5 mg film coated tablet and placebo for saxagliptin as an add-on to metformin (≥1500 mg/day orally)
- Saxagliptin + Metformin: Randomized participants received orally QD saxagliptin 5 mg film coated tablet and placebo for dapagliflozin as an add-on to metformin (≥1500 mg/day orally)
Period: 1 -Modified Enrolled Participants Set
Arm/Group | Dapagliflozin + Saxagliptin + Metformin | Dapagliflozin + Metformin | Saxagliptin + Metformin
Started (7 participants of 1 US site were excluded due to serious Good Clinical Practice (GCP)) | 293 | 294 (A participant was randomized but did not receive treatment) | 296 (A participant was randomized but did not receive treatment)
Participants Completed Treatment Period | 273 | 276 | 283
Completed (Participants who completed study treatment) | 256 | 255 | 243
Not Completed | 37 | 39 | 53
Not completed — Participant decision | 7 | 10 | 9
Not completed — Adverse Event | 10 | 4 | 1
Not completed — Severe non-compliance to protocol | 2 | 0 | 1
Not completed — Lack of therapeutic response | 1 | 5 | 14
Not completed — Study-specific discontinuation criteria | 11 | 13 | 20
Not completed — Other | 6 | 6 | 7
Not completed — No treatment given | 0 | 1 | 1
Period: 2 - Enrolled Participants Set
Arm/Group | Dapagliflozin + Saxagliptin + Metformin | Dapagliflozin + Metformin | Saxagliptin + Metformin
Started (Includes 7 participants of one US site which was excluded in Modified Enrolled participants set) | 301 (Population was used for the sensitivity analysis to assess the robustness of the treatment effect.) | 302 (Population was used for the sensitivity analysis to assess the robustness of the treatment effect.) | 302 (Population was used for the sensitivity analysis to assess the robustness of the treatment effect.)
Participants Completed Treatment Period | 281 | 284 (A participant was randomized but did not receive treatment due to screen failure.) | 289 (A participant was randomized but did not receive treatment due to screen failure.)
Completed (Participants who completed study treatment) | 261 | 261 | 248
Not Completed | 40 | 41 | 54
Not completed — Participant decision | 7 | 10 | 9
Not completed — Adverse Event | 10 | 4 | 1
Not completed — Severe non-compliance to protocol | 2 | 0 | 1
Not completed — Lack of therapeutic response | 1 | 5 | 14
Not completed — Study specific discontinuation criteria | 14 | 15 | 21
Not completed — Other | 6 | 6 | 7
Not completed — No treatment given | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): All randomized participants who took at least 1 dose of study drug & had baseline value for HbA1c. Analysis was based on randomized treatment. Modified FAS - all participants from FAS with the exception of participants from one site (United States; excluded due to serious Good Clinical Practice [GCP] violations).
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin + Saxagliptin + Metformin | Dapagliflozin + Metformin | Saxagliptin + Metformin | Total
Number analyzed (Participants) | 290 | 289 | 291 | 870
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.2 (10.68) | 55.9 (10.94) | 57.0 (9.94) | 56.7 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 137 | 134 | 419
  Male | 142 | 152 | 157 | 451
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 99 | 95 | 99 | 293
  Not Hispanic or Latino | 191 | 194 | 192 | 577
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 0 | 4
  Asian | 9 | 9 | 6 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 17 | 24 | 51
  White | 265 | 257 | 258 | 780
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 3 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at Week 24
Description: To demonstrate the superiority of the change from baseline HbA1c achieved with the co-administered saxagliptin 5 mg and dapagliflozin 5 mg to either agent individually after 24 weeks. Results were presented for the modified full analysis set.
  Note: Baseline was defined as the last assessment on or prior to the date of the first dose of the study medication.
Time Frame: Baseline and week 24
Population: FAS: All randomized participants who took at least one dose of the study medication and had a baseline value for HbA1c. Analysis of the FAS was based on the randomized treatment. The modified FAS included all participants from FAS with the exception of participants from one site (excluded due to serious GCP violations).
Measure: Least Squares Mean (Standard Error); unit: Percentage (%)
Arm/Group | Dapagliflozin + Saxagliptin + Metformin | Dapagliflozin + Metformin | Saxagliptin + Metformin
Number analyzed (Participants) | 290 | 289 | 291
Percentage (%) | -1.03 (0.0558) | -0.63 (0.0560) | -0.69 (0.0551)
Statistical Analysis 1: Comparison: Dapagliflozin + Saxagliptin + Metformin vs Dapagliflozin + Metformin; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -0.40, 95% CI 2-sided [-0.55 to -0.24]
Statistical Analysis 2: Comparison: Dapagliflozin + Saxagliptin + Metformin vs Saxagliptin + Metformin; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -0.34, 95% CI 2-sided [-0.50 to -0.19]

2. Secondary Outcome: Proportion of Participants Achieving HbA1c <7.0% at 24 Weeks
Description: To demonstrate the effect of the co-administered saxagliptin 5 mg and dapagliflozin 5 mg to either agent individually on proportion of participants achieving therapeutic glycaemic response after 24 weeks. Therapeutic glycaemic response was defined as an HbA1c value at Week 24 <7.0% irrespective of whether participant received rescue medication. Risk difference for each treatment was calculated as adjusted response rate. Participants who did not had an HbA1c measurement at Week 24 were regarded as non-responders. Results were presented for the modified full analysis set.
Time Frame: Baseline and week 24
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Dapagliflozin + Saxagliptin + Metformin | Dapagliflozin + Metformin | Saxagliptin + Metformin
Number analyzed (Participants) | 290 | 289 | 291
Participants | 124 | 63 | 83
Statistical Analysis 1: Comparison: Dapagliflozin + Saxagliptin + Metformin vs Dapagliflozin + Metformin; Test type: Superiority; p < 0.0001, Method of Zhang, Tsiatis, and Davidian; Risk Difference (RD) = 19.8, 95% CI 2-sided [12.7 to 26.9]
Statistical Analysis 2: Comparison: Dapagliflozin + Saxagliptin + Metformin vs Saxagliptin + Metformin; Test type: Superiority; p = 0.0018, Method of Zhang, Tsiatis, and Davidian; Risk Difference (RD) = 11.7, 95% CI 2-sided [4.4 to 19.1]

3. Secondary Outcome: Change in Fasting Plasma Glucose at 24 Weeks
Description: To demonstrate the effect of the co-administered saxagliptin 5 mg and dapagliflozin 5mg to either agent individually on fasting plasma glucose after 24 weeks. Results were presented for the modified full analysis set.
Time Frame: Baseline and week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Milligrams per deciliter (mg/dL)
Arm/Group | Dapagliflozin + Saxagliptin + Metformin | Dapagliflozin + Metformin | Saxagliptin + Metformin
Number analyzed (Participants) | 290 | 289 | 291
Milligrams per deciliter (mg/dL) | -27.53 (2.1557) | -19.95 (2.1738) | -12.66 (2.1373)
Statistical Analysis 1: Comparison: Dapagliflozin + Saxagliptin + Metformin vs Dapagliflozin + Metformin; Test type: Superiority; p = 0.0135, Mixed Models Analysis; LS mean difference = -7.58, 95% CI 2-sided [-13.59 to -1.57]
Statistical Analysis 2: Comparison: Dapagliflozin + Saxagliptin + Metformin vs Saxagliptin + Metformin; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -14.88, 95% CI 2-sided [-20.85 to -8.91]

4. Secondary Outcome: Change in Total Body Weight at 24 Weeks
Description: To demonstrate the effect of the co-administered saxagliptin 5 mg and dapagliflozin 5 mg to saxagliptin 5 mg on total body weight after 24 weeks. Results were presented for the modified full analysis set.
Time Frame: Baseline and week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Kilograms (Kg)
Arm/Group | Dapagliflozin + Saxagliptin + Metformin | Saxagliptin + Metformin
Number analyzed (Participants) | 290 | 291
Kilograms (Kg) | -2.01 (0.1829) | -0.41 (0.1815)
Statistical Analysis 1: Comparison: Dapagliflozin + Saxagliptin + Metformin vs Saxagliptin + Metformin; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.60, 95% CI 2-sided [-2.11 to -1.09]

ADVERSE EVENTS:
Time Frame: From time of randomization, and throughout the treatment period and until end of treatment (Visit 5)/early termination + 4 days for non serious AEs and 30 days for SAEs.
Description: An undesirable medical condition could be symptoms (eg, nausea, chest pain), signs (eg, tachycardia, enlarged liver)/abnormal results of an investigation (eg, laboratory findings, electrocardiogram). One participant was randomized but did not receive treatment in Dapagliflozin+Metformin and Saxagliptin + Metformin groups.
Arm/Group | Dapagliflozin + Saxagliptin + Metformin | Dapagliflozin + Metformin | Saxagliptin + Metformin
All-Cause Mortality (participants affected / at risk) | 1/293 | 2/293 | 0/295
Serious Adverse Events (participants affected / at risk) | 7/293 | 8/293 | 7/295
Other Adverse Events (participants affected / at risk) | 41/293 | 39/293 | 29/295
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin + Saxagliptin + Metformin (N=293) | Dapagliflozin + Metformin (N=293) | Saxagliptin + Metformin (N=295)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Basal ganglia haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arteritis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin + Saxagliptin + Metformin (N=293) | Dapagliflozin + Metformin (N=293) | Saxagliptin + Metformin (N=295)
Glomerular filtration rate decreased (Investigations) | 12 (13) | 11 (11) | 5 (5)
Urinary tract infection (Infections and infestations) | 7 (7) | 3 (4) | 5 (5)
Pollakiuria (Renal and urinary disorders) | 7 (8) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 5 (5) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 5 (5) | 9 (10) | 8 (8)
Influenza (Infections and infestations) | 3 (3) | 9 (9) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 4 (4) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All clinical study findings and documents will be regarded as confidential. The investigator and members of his/her research team must not disclose such information without prior written approval from the sponsor.

DOCUMENTS (2):
  • Study Protocol (2016-08-04): https://cdn.clinicaltrials.gov/large-docs/94/NCT02681094/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT02681094/SAP_001.pdf